CLINICAL TRIAL: NCT01005329
Title: A Phase II Study of Postoperative Intensity Modulated Radiation Therapy (IMRT) With Concurrent Cisplatin and Bevacizumab Followed by Carboplatin and Paclitaxel for Patients With Endometrial Cancer
Brief Title: Intensity-Modulated Radiation Therapy, Cisplatin, and Bevacizumab Followed by Carboplatin and Paclitaxel in Treating Patients Who Have Undergone Surgery for Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01982; NCI-2011-01982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000657979; RTOG-0921; RTOG 0921 (Other: Radiation Therapy Oncology Group); RTOG-0921 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Stage IA Uterine Corpus Cancer AJCC v7; Stage IB Uterine Corpus Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes

ARMS (1):
- Treatment (IMRT, cisplatin,bevacizumab,carboplatin,paclitaxel) (Experimental): Patients undergo pelvic IMRT once daily, 5 days a week, for 5 weeks. Patients may also undergo optional nodal boost radiotherapy and/or vaginal brachytherapy boost. Patients also receive concurrent cisplatin IV over 1 hour on days 1 and 29 and bevacizumab IV over 30-90 minutes on days 1, 15, and 29. Beginning 4-6 weeks after completing IMRT, cisplatin, and bevacizumab, patients receive carboplatin IV over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment with carboplatin and paclitaxel repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Drug: Paclitaxel

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial studies the side effects of giving intensity-modulated radiation therapy together with cisplatin and bevacizumab followed by carboplatin and cisplatin and to see how well they work in treating patients who have undergone surgery for high-risk endometrial cancer. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin, carboplatin, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving intensity-modulated radiation therapy together with chemotherapy and bevacizumab after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the treatment-related, grade 3+, non-hematologic adverse-event rate within 90 days from the start of treatment with concurrent intensity-modulated radiotherapy, cisplatin, and bevacizumab followed by carboplatin and paclitaxel in patients with high-risk endometrial cancer.

SECONDARY OBJECTIVES:

I. To evaluate treatment-related adverse events occurring within 1 year from the start of treatment.

II. To evaluate all treatment-related adverse events. III. To evaluate disease-free and overall survival. IV. To evaluate local, regional, and distant failure.

OUTLINE:

Patients undergo pelvic intensity-modulated radiotherapy (IMRT) once daily, 5 days a week, for 5 weeks. Patients may also undergo optional nodal boost radiotherapy and/or vaginal brachytherapy boost. Patients also receive concurrent cisplatin intravenously (IV) over 1 hour on days 1 and 29 and bevacizumab IV over 30-90 minutes on days 1, 15, and 29. Beginning 4-6 weeks after completing IMRT, cisplatin, and bevacizumab, patients receive carboplatin IV over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment with carboplatin and paclitaxel repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer, including 1 of the following cellular types:

  * Endometrioid endometrial adenocarcinoma
  * Clear cell carcinoma
  * Papillary serous adenocarcinoma
  * Adenosquamous cell carcinoma
  * Other adenocarcinoma variant
* No carcinosarcoma
* Meets 1 of the following criteria:

  * Grade 3 carcinoma with > 50% myometrial invasion (stage IC or IIA) (all papillary serous or clear cell carcinoma will be considered grade 3)
  * Grade 2 or 3 carcinoma with any cervical stromal invasion (stage IIB)
  * Known extra-uterine disease confined to the pelvis (stage III or IVA)

    * Patients with stage III or IVA disease must have undergone computed tomography (CT) scan or positron emission tomography (PET)/CT scan of the abdomen and pelvis within the past 56 days
* Has undergone hysterectomy (i.e., total abdominal, vaginal, robotic-assisted, radical, or laparoscopic-assisted vaginal hysterectomy) and bilateral salpingo-oophorectomy within the past 56 days
* No positive common iliac or positive para-aortic nodal disease (defined as lymph nodes ? 2 cm in any dimension on CT scan or biopsy) or positive peritoneal cytology
* No evidence of metastatic extrauterine disease, gross or residual disease (not including pelvic nodal disease), or distant metastases
* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ? 1,500/mm^3 (without growth factor support)
* Platelet count ? 100,000/mm^3
* Hemoglobin ? 10 g/dL (transfusion allowed)
* Total bilirubin ? 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ? 2 times ULN
* Serum creatinine ? 1.5 mg/dL
* Urine protein:creatinine ratio ? 0.5 OR urine protein < 1,000 mg on 24-hour urine collection
* International normalized ratio (INR) < 1.5 (for patients treated with warfarin within the past 14 days)
* Not nursing
* No neuropathy ? Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* No ototoxicity > CTCAE grade 2
* No serious, active comorbidity, including any of the following:

  * Unstable angina and/or New York Heart Association (NYHA) class II-IV congestive heart failure requiring hospitalization within the past 12 months
  * Transmural myocardial infarction within the past 12 months
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control (CDC) definition (human immunodeficiency virus [HIV] testing is not required)
  * Active gastrointestinal (GI) ulcers, GI bleeding, inflammatory bowel disease, or GI obstruction
  * Inadequately controlled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg and/or diastolic BP > 90 mm Hg on antihypertensive medications
  * Significant vascular disease, including aortic aneurysm, aortic dissection, or arteriovenous malformation within the past 12 months
  * Serious cardiac arrhythmia on medication (well-controlled atrial fibrillation on medication allowed)
  * Serious non-healing wound, ulcer, or bone fracture
* No history of hypertensive crisis or hypertensive encephalopathy
* No stroke/cerebrovascular event within the past 12 months
* No arterial thromboembolic events, including transient ischemic attack or clinically symptomatic peripheral artery disease within the past 12 months
* No abdominal fistula, GI perforation, or intra-abdominal abscess within the past 6 months
* No other invasive malignancies within the past 3 years other than nonmelanomatous skin cancer
* No significant trauma within the past 28 days
* No mental status changes or bladder problems that would preclude the ability to comply with bladder-filling instructions
* No mental or psychiatric illness that would preclude giving informed consent
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No prior allergic reaction to bevacizumab, cisplatin, carboplatin, or paclitaxel
* No concurrent erythropoietin, St. John's wort, therapeutic anticoagulants, aminoglycoside antibiotics, or amifostine
* No prior organ transplantation
* No prior external-beam radiotherapy to the pelvis resulting in overlapping of radiotherapy fields
* No prior systemic chemotherapy for uterine cancer

  * Prior chemotherapy for a different cancer is allowed
* No prior therapy with anti-vascular endothelial growth factor (VEGF) compounds
* More than 28 days since prior major surgical procedure requiring open biopsy incision
* No concurrent surgery (except for vascular access device placement or procedures that do not require significant incision)
* No concurrent warfarin at doses > 1 mg/day

  * Concurrent prophylactic low molecular weight heparin allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11-06 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2013-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akila Viswanathan, Principal Investigator — Radiation Therapy Oncology Group
Locations (41):
- United States (38):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Bay Medical Center, Panama City, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Elliot Hospital, Manchester, New Hampshire
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - London Regional Cancer Program, London, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong

REFERENCES:
- [Result] Viswanathan AN, Moughan J, Miller BE, Xiao Y, Jhingran A, Portelance L, Bosch WR, Matulonis UA, Horowitz NS, Mannel RS, Souhami L, Erickson BA, Winter KA, Small W Jr, Gaffney DK. NRG Oncology/RTOG 0921: A phase 2 study of postoperative intensity-modulated radiotherapy with concurrent cisplatin and bevacizumab followed by carboplatin and paclitaxel for patients with endometrial cancer. Cancer. 2015 Jul 1;121(13):2156-63. doi: 10.1002/cncr.29337. Epub 2015 Apr 6. PMID 25847373

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation (IMRT), Chemotherapy: Pelvic intensity-modulated radiation therapy (IMRT) once daily, 5 days a week, for 5 weeks (45 Gy in 25 fractions) with optional nodal boost radiotherapy and/or vaginal brachytherapy boost. Concurrent cisplatin (CISPT) 50 mg/m^2 IV over 1 hour on days 1 and 29 and bevacizumab (BEV) 5mg/kg IV over 30-90 minutes on days 1, 15, and 29. Beginning 4-6 weeks after completing IMRT, cisplatin, and bevacizumab, patients receive carboplatin (CBCDA) IV area under the curve (AUC) 5 over 1 hour and paclitaxel (PTX) IV 135 mg/m^2 over 3 hours on day 1 and every every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Started | 34
Completed | 30 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 4
Not completed — Ineligible or received no protocol trt. | 4

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Chemoradiation (IMRT), Chemotherapy: Pelvic intensity-modulated radiation therapy (IMRT) once daily, 5 days a week, for 5 weeks (45 Gy in 25 fractions) with optional nodal boost radiotherapy and/or vaginal brachytherapy boost. Concurrent cisplatin (CISPT) 50 mg/m^2 IV over 1 hour on days 1 and 29 and bevacizumab (BEV) 5mg/kg IV over 30-90 minutes on days 1, 15, and 29. Beginning 4-6 weeks after completing IMRT, cisplatin, and bevacizumab, patients receive carboplatin (CBCDA) IV AUC 5 over 1 hour and paclitaxel (PTX) IV 135 mg/m^2 over 3 hours on day 1 and every every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-related, Grade 3+, Non-hematologic Adverse Events Occuring Within 90 Days After Treatment Start
Description: Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE, assigning Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to 90 days
Population: Eligible patients who started study treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 23.3 [10.63 to 36.0]
Statistical Analysis 1: Comparison: Chemoradiation (IMRT), Chemotherapy; Test type: Other; The rate of the acute specified AEs (adverse events) from previous (and prior to ClinicalTrials.gov requirements) Radiation Therapy Oncology Group (RTOG) trial 9708 of RT + cisplatin was 44% and the hypothesis is that the addition of bevacizumab to IMRT + cisplatin will not increase this rate beyond 60%. This study was designed with a 1-sided, upper bound confidence interval to estimate this AE rate. Twenty-seven evaluable patients were required to have 95% confidence that the true grade 3+ non-hematologic treatment-related AE rate is not greater than 60%. Please note that this is a 95% ONE-SIDED confidence bound which is equivalent to the upper bound of a two-sided 90% confidence interval

2. Secondary Outcome: Percentage of Participants With Treatment-related, Grade 3+, Non-hematologic Adverse Events Occuring Within 1 Year After Treatment Start
Description: Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE, assigning Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Adverse events reported as definitely, probably, or possibly related to study treatment.
Time Frame: From start of treatment to one year
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 43.3 [28.5 to 58.2]

3. Secondary Outcome: Treatment-related Grade 3+ Adverse Events
Description: The highest grade adverse event per patient reported as definitely, probably, or possibly related to study treatment is counted. Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE, assigning Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to end of follow-up, up to 43.4 months; analysis occurred after all patients had been on study for at least one year.
Population: Eligible patients who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
Participants
  Grade 0 | 1
  Grade 1 | 0
  Grade 2 | 8
  Grade 3 | 12
  Grade 4 | 9
  Grade 5 | 0

4. Secondary Outcome: Overall Survival (Two-year Rate Reported)
Description: Failure was defined as death due to any cause. Patients alive at time of analysis were censored at the date of last contact. Survival rate at two years was estimated using the Kaplan-Meier method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 96.7 [78.6 to 99.5]

5. Secondary Outcome: Disease-free Survival (Two-year Rate Reported)
Description: Failure was defined as pelvic failure (recurrence in the pelvis, which must be confirmed by histologic or cytologic biopsy of the recurrent lesion), distant failure (confirmed by histologic or cytologic biopsy of the recurrent lesion), or death due to any cause. Patients alive at time of analysis were censored at the date of last contact. Disease-free survival rate at two years was estimated using the Kaplan-Meier method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 79.1 [59.2 to 90.1]

6. Secondary Outcome: Pelvic Failure Rate (Two-year Rate Reported)
Description: Pelvic failure (PF) was defined as disease recurrence in the pelvis, including the pelvic or sacral lymph nodes, and required confirmation by histologic or cytologic biopsy of the recurrent lesion. Death was considered a competing risk. PF rates were estimated using the cumulative incidence method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 0 [0 to 0]

7. Secondary Outcome: Distant Failure (Two-year Rate Reported)
Description: Distant Failure (DF) was defined as the appearance of distant metastasis. Death was considered a competing risk. DF rates were estimated using the cumulative incidence method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Number analyzed (Participants) | 30
percentage of participants | 17.0 [3.2 to 30.9]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Arm/Group | Chemoradiation (IMRT), Chemotherapy
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation (IMRT), Chemotherapy (N=30)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Neuralgia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation (IMRT), Chemotherapy (N=30)
Anemia (Blood and lymphatic system disorders) | 22
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 5
Blurred vision (Eye disorders) | 8
Eye disorders - Other, specify (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Anal mucositis (Gastrointestinal disorders) | 1
Anal pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 18
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 22
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 19
Proctitis (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 4
Rectal pain (Gastrointestinal disorders) | 3
Salivary duct inflammation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Chills (General disorders) | 3
Edema face (General disorders) | 2
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 26
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 3
Localized edema (General disorders) | 1
Pain (General disorders) | 5
Bladder infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urethral infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Vaginal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 5
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 5
GGT increased (Investigations) | 2
Hemoglobin increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 6
Lymphocyte count decreased (Investigations) | 19
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 16
Weight gain (Investigations) | 2
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 23
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 14
Syncope (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5
Urinary frequency (Renal and urinary disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 8
Urinary urgency (Renal and urinary disorders) | 5
Breast pain (Reproductive system and breast disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 6
Vaginal dryness (Reproductive system and breast disorders) | 7
Vaginal hemorrhage (Reproductive system and breast disorders) | 4
Vaginal inflammation (Reproductive system and breast disorders) | 3
Vaginal pain (Reproductive system and breast disorders) | 3
Vaginal stricture (Reproductive system and breast disorders) | 3
Vaginismus (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 17
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 3
Hot flashes (Vascular disorders) | 8
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less